CLINICAL TRIAL: NCT02272218
Title: Bariatric Lap Band Surgery as a Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-03313
Record Dates: First submitted 2014-10-10; First posted 2014-10-22 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAGB (Other): There is only one arm for this study, since this study involves a single cohort receiving the same intervention, laparoscopic gastric banding (LAGB) surgery.
  Interventions: Procedure: bariatric lap band surgery

INTERVENTIONS:
Procedure: bariatric lap band surgery — The intervention in this study is laparoscopic gastric banding (LAGB) surgery as a treatment option for obese patients with pain from knee osteoarthritis (KOA) refractory to medical treatment

SUMMARY:
The primary purpose of this study is to evaluate laparoscopic gastric banding (LAGB) surgery as a treatment option for obese patients with pain from knee osteoarthritis (KOA) refractory to medical treatment. The primary outcome will be the reduction in OA-related pain and disability after LAGB.

DETAILED DESCRIPTION:
This is a pilot study of 15 (may need to consent/screen 30 patients to have 15 enrolled) obese patients (BMI 30-40) with painful knee osteoarthritis. Although prior studies have reported musculoskeletal secondary outcomes following various types of bariatric surgery, investigators propose the evaluation of laparoscopic gastric banding (LAGB) to treat a cohort of patients with moderate to severe knee osteoarthritis.

Once eligible patients are identified by rheumatologists and/or bariatric team and consented for the study, they will have bilateral knee radiographs (standard of care) to ensure they have a sufficient degree of OA. Patients will then be referred to the bariatric surgeons, who will then confirm the patients' interest, understanding and suitability for the LAGB surgery which is a FDA approved procedurefor patients with a BMI >30 and at least one obesity-related comorbidity (including knee OA)37. It is the application of this approved procedure that constitutes the research question should LAGB surgery be considered as a treatment option to improve pain and physical disability in patients with knee OA? During the pre-operative process patients will be given study questionnaires to evaluate knee pain and function, have a musculoskeletal exam and blood/urine will be collected.These procedures will be repeated at post-operative intervals to track response of the knees to the LAGB.

The primary outcome measure is improvement in OA-related knee pain and physical disability. Improvement of pain and function will be defined by changes in the VAS, WOMAC, AORC and KOOS scores. The degree of improvement required to qualify as such will be described in the methods sections below.

Secondary outcome measures include (1) radiographic evidence of OA progression or worsening despite the LABG, (2) weight loss, and (3) reduction or discontinuation of pain medication.

ELIGIBILITY:
Inclusion Criteria:

1. able and willing to provide written informed consent
2. at least 25 years of age
3. body mass index (BMI) between 30 and 40 (FDA-approved BMI window for LAGB surgery if there is at least one comorbidity)
4. pain in at least one knee for 15 of the 30 days prior to screening

   1. clinically diagnosed with knee OA using American College of Rheumatology (ACR) criteria.
   2. Patient pain visual analog scale (VAS) ≥40
   3. pain not controlled with Tylenol, NSAIDs or topical therapy (or unable to use/tolerate NSAIDs for medical reasons)
5. anterior-posterior (AP) radiograph of at least one knee with Kellgren-Lawrence (K-L) grading scale ≥ 2 (moderate to severe osteoarthritis)

Exclusion Criteria:

1. unable to provide written informed consent
2. less than 25 yrs of age
3. BMI <30 or >40
4. does not fulfill the ACR criteria for OA
5. VAS <40
6. any clinical disorder requiring use of corticosteroids within one week of visit
7. viscosupplementation or intra-articular steroid injection to the affected knee within the prior one month
8. bilateral total knee replacement
9. has not yet tried to treat pain with oral NSAIDs/COX-2 inhibitors (unless medical contraindications), Tylenol, or topical therapy
10. co-morbidities including, congestive heart failure, hepatic or renal disease, chronic infectious diseases, non-cutaneous cancer within last five years
11. comorbidities that would make lap band surgery contraindicated (severe cardiopulmonary diseases, severe esophagitis, stomach or duodenal ulcers, esophageal or gastric varices, inflammatory bowel disease, liver cirrhosis, chronic pancreatitis, alcohol or drug addiction, on chronic steroid treatment, or active infections)
12. anterior-posterior (AP) radiograph of both knees with K-L grade < 2
13. pregnancy or women of childbearing potential with a positive pregnancy test during pre-surgical phases of the study as part of standard of care pre-op testing.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
reduction in OA-related pain and disability after LAGB. | 4 years
  questionnaires will be distributed pre- and post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Musculoskeletal Care, New York, New York, United States